CLINICAL TRIAL: NCT02153905
Title: A Phase I-II Study of the Treatment of Metastatic Cancer That Expresses MAGE-A3 Using Lymphodepleting Conditioning Followed by Infusion of Anti-MAGE-A3 HLA-A*01 Restricted TCR-Gene Engineered Lymphocytes and Aldesleukin
Brief Title: T Cell Receptor Immunotherapy Targeting MAGE-A3 for Patients With Metastatic Cancer Who Are HLA-A*01 Positive
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow, insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 140110; 14-C-0110
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer; Cervical Cancer; Renal Cancer; Melanoma; Bladder Cancer
Keywords: Melanoma; Immunotherapy; Metastatic Cancer; Gene Therapy; T Cells
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Kidney Neoplasms; Melanoma; Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — aldesleukin; Interleukin-2; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 - Dose Escalation/De-Escalation (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MAGE-A3- A1 transduced peripheral blood lymphocytes (PBL) + high-dose aldesleukin
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-MAGE-A3 human leukocyte antigen serotype within HLA-A A serotype group (HLA-A* 01)-restricted T-cell receptor (TCR)
- Phase II - Maximum Tolerated Dose (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MAGE-A3- A1 transduced peripheral blood lymphocytes (PBL) + high-dose aldesleukin
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-MAGE-A3 human leukocyte antigen serotype within HLA-A A serotype group (HLA-A* 01)-restricted T-cell receptor (TCR)

INTERVENTIONS:
Drug: Aldesleukin — Aldeskeukin 720,000 IU/kg (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Other Names: Interleukin-2
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Other Names: Cytoxan
Biological: Anti-MAGE-A3 human leukocyte antigen serotype within HLA-A A serotype group (HLA-A* 01)-restricted T-cell receptor (TCR) — Day 0: MAGE-A3-A1 transduced peripheral blood lymphocytes (PBL) will be infused intravenously on the Patient Care Unit over 20-30 minutes.

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patients white blood cells with a retrovirus that has the gene for anti-MAGE-A3 incorporated in the retrovirus.

Objective:

The purpose of this study is to determine a safe number of these cells to infuse and to see if these particular tumor-fighting cells (anti-MAGE A3 cells) cause tumors to shrink and to be certain the treatment is safe

Eligibility:

- Adults age 18-66 with cancer expressing the MAGE-A3 molecule.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti MAGE-A3 cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti MAGE-A3 cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains both alpha and beta chains of a T cell receptor (TCR) that recognizes the human leukocyte antigen serotype within HLA-A "A" serotype group (HLA-A 01) restricted MAGE-A3 tumor antigen, which can be used to mediate genetic transfer of this TCR with high efficiency.
* In co-cultures with human leukocyte antigen serotype within HLA-A A serotype group (HLA-A 01) and MAGE-A3 double positive tumors, the anti-MAGE-A3- A 01 restricted (anti-MAGE-A3-01) TCR transduced T cells secreted significant amounts of Interferon (IFN)- >= with high specificity.

Objectives:

Primary objectives:

* Determine a safe dose of administration of autologous T cells transduced with an anti- MAGE-A3 HLA-A 01-restricted TCR (MAGE-A3-01) TCR and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen.
* Determine if this approach will result in objective tumor regression in patients with metastatic cancer expressing MAGE-A3.
* Determine the toxicity profile of this treatment regimen.

Eligibility:

Patients who are HLA-A 01 positive and 18 years of age or older must have

* Metastatic cancer whose tumors express the MAGE-A3 antigen
* Previously received and have been a non-responder to or recurred following at least one first line treatment for metastatic disease

Patients may not have:

- Contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis will be transduced with the retroviral vector supernatant encoding the anti-MAGE-A3 HLA-A 01-restricted TCR.
* The study will begin with a phase I dose escalation. After the maximum tolerated dose (MTD) cell dose has been determined, patients will be enrolled into the phase II portion of the trial at the MTD established during the phase I portion of the study. In the phase II portion, patients will be entered into two cohorts: cohort 2a will include patients with metastatic melanoma; cohort 2b will include patients with renal cancer and other types of metastatic cancer.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene-transduced PBMC plus intravenous (IV) aldesleukin.
* Patients will undergo complete evaluation of tumor response every 1-6 months until off study criteria are met.
* For each of the two strata evaluated in the phase 2 portion, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* For both strata, the objective will be to determine if the treatment regimen is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modes 20% partial response (PR) + complete response (CR) rate (p1=0.20).
* In order to complete the dose escalation phase and both phase II cohorts, a total of up to 20+82=102 patients may be required (20 + 2 strata with a maximum of 41 apiece). Up to 6 patients enrolled at the MTD will count towards the accrual in the appropriate phase II strata if they are evaluable for response and if they would be fully eligible for enrollment in the phase II portion of the trial. Provided that about 4-5 patients per month will be able to be enrolled onto this trial, approximately 2 to 3 years may be needed to accrue the maximum number of required patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic or locally advanced refractory/recurrent cancer that expresses MAGE-A3 as assessed by one of the following methods: reverse transcription polymerase chain reaction (RT-PCR) on tumor tissue defined as 30,000 copies of MAGE-A3 per 106 glyceraldehyde 3-phosphate dehydrogenase (GAPDH) copies, or by immunohistochemistry of resected tissue defined as 10% or greater of tumor cells being 2-3+ for MAGE-A3, or serum antibody reactive with MAGE-A3. Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the National Cancer Institute (NCI).
  2. Patients must have previously received prior first line standard therapy (or effective salvage chemotherapy regimens) for their disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
  3. Patients must be human leukocyte antigen serotype within HLA-A A serotype group (HLA-A*01) positive.
  4. Greater than or equal to 18 years of age and less than or equal to age 70.
  5. Ability of subject to understand and the willingness to sign the Informed Consent Document
  6. Willing to sign a durable power of attorney
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1
  8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
  9. Serology:

     * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
  10. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
  11. Hematology

      * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
      * White blood cell (WBC) greater than or equal to 3000/mm^3
      * Platelet count greater than or equal to 100,000/mm^3
      * Hemoglobin > 8.0 g/dl
  12. Chemistry:

      * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to to 2.5 times the upper limit of normal
      * Serum creatinine less than or equal to to 1.6 mg/dl
      * Total bilirubin less than or equal to to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  13. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients must have progressing disease after prior treatment. Note: Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies
  14. Subjects must be co-enrolled in protocol 03-C-0277.

Note: Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Active systemic infections (e.g.: requiring anti-infective treatment), coagulation disorders or any other active major medical illnesses.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of any cardiac events including coronary revascularization or ischemic symptoms.
8. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45%; testing is required in patients who are:

   * Age greater than or equal to 65 years old
   * Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or have a history of ischemic heart disease, or chest pain.
9. Patients with central nervous system (CNS) metastases or symptomatic CNS involvement (including cranial neuropathies or mass lesions).
10. Patients presenting with lesions that may harbor an occult infectious source.
11. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
    * Symptoms of respiratory dysfunction
12. Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07-03 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan RA, Dudley ME, Yu YY, Zheng Z, Robbins PF, Theoret MR, Wunderlich JR, Hughes MS, Restifo NP, Rosenberg SA. High efficiency TCR gene transfer into primary human lymphocytes affords avid recognition of melanoma tumor antigen glycoprotein 100 and does not alter the recognition of autologous melanoma antigens. J Immunol. 2003 Sep 15;171(6):3287-95. doi: 10.4049/jimmunol.171.6.3287. PMID 12960359
- [Background] Johnson LA, Morgan RA, Dudley ME, Cassard L, Yang JC, Hughes MS, Kammula US, Royal RE, Sherry RM, Wunderlich JR, Lee CC, Restifo NP, Schwarz SL, Cogdill AP, Bishop RJ, Kim H, Brewer CC, Rudy SF, VanWaes C, Davis JL, Mathur A, Ripley RT, Nathan DA, Laurencot CM, Rosenberg SA. Gene therapy with human and mouse T-cell receptors mediates cancer regression and targets normal tissues expressing cognate antigen. Blood. 2009 Jul 16;114(3):535-46. doi: 10.1182/blood-2009-03-211714. Epub 2009 May 18. PMID 19451549
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The two groups below represent the Phase I period. Study was terminated prior to the phase II portion due to slow, insufficient accrual.
Groups:
- Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2); Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MAGE-A3- A1 transduced peripheral blood lymphocytes (PBL) + high-dose aldesleukin
  Aldesleukin: Aldeskeukin 720,000 IU/kg (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Fludarabine: Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Cyclophosphamide: Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Anti-MAGE-A3 human leukocyte antigen serotype within HLA-A A serotype group (HLA-A* 01)-restricted T-cell receptor (TCR): Day 0: MAGE-A3-A1 transduced peripheral blood lymphocytes (PBL) will be infused intravenously on the Patient Care Unit over 20-30 minutes.
Period: Overall Study
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Started | 1 | 2
Completed | 0 | 2
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (0) | 50.8 (11.88) | 53 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Cell Dose (MTD)
Description: Highest dose at which less than or equal to 1 of 6 patients experienced a dose limiting toxicity (DLT) or the highest dose level studied if DLTs are not observed at any of the dose levels. DLT is defined as follows: Grade 3-5 allergic reactions related to the study cell infusion. Grade 3 and greater autoimmune reactions. Grades 3 and greater organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to the underlying malignancy and occurring within 30 days of study cell infusion and does not resolve within 72 hours. Treatment-related death within 8 weeks of the study cell infusion.
Time Frame: Within 30 days of study cell infusion, before progression to next-higher dose level
Population: The first participant in the first Arm/Group experienced a dose limiting toxicity so the second cohort was a de-escalation and was not completed. As a result, maximum tolerated dose was not determined.
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Patients With Objective Tumor Regression
Description: Objective tumor regression is defined as the number of participants with a complete or partial response per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 6 and 12 weeks after cell infusion on up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Number analyzed (Participants) | 1 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1

3. Primary Outcome: Number of Treatment Related Adverse Events Related to T-Cell Receptor (TCR) Gene-Engineered Cells
Description: Aggregate of all Grade ≥3 adverse events and their frequency possibly, probably or definitely related to the research. Adverse Events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v.4.0. Grade 3 is severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL). Grade 4 is life-threatening consequences; urgent intervention indicated. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to end of treatment, approximately 30 days
Measure: Number; unit: adverse events
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Number analyzed (Participants) | 1 | 2
adverse events
  Grade 3 Atrial Fibrillation | 1 | 0
  Grade 3 Diarrhea | 1 | 0
  Grade 3 Ileus | 1 | 0
  Grade 3 Edema face: anasarca | 1 | 0
  Grade 3 Fibrinogen decreased | 1 | 0
  Grade 3 aPTT prolonged | 1 | 0
  Grade 3 Acute Kidney Injury | 1 | 0
  Grade 3 Rash maculo-papular | 1 | 0
  Grade 4 Hemophagocytic Syndrome | 1 | 0
  Grade 4 Blood bilirubin increased | 1 | 0
  Grade 4 Depressed level of consciousness | 1 | 0
  Grade 4 Encephalopathy | 1 | 0
  Grade 4 Hypotension | 1 | 0

4. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 53 days for the Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) Arm/Group, and 1 year and 4 months for the Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2) Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

5. Secondary Outcome: In Vivo Survival of T-Cell Receptor (TCR) Cells
Description: In vivo survival of gene-engineered lymphocytes derived from the infused cells will be analyzed by tetramer analysis and staining for the T-cell receptor (TCR). Tetramer analysis is measured by % of peripheral blood.
Time Frame: Up to 3 years after study cell infusion
Population: Data is not reported due to dose limiting toxicities leading to premature stop of dose escalation, and also lack of durable objective tumor regression demonstrated by all three patients. Because no further resources will be expended on this closed study, analysis of this secondary outcome measure (via tetramer analysis) will not be performed.
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT is defined as follows: Grade 3-5 allergic reactions related to the study cell infusion. Grade 3 and greater autoimmune reactions. Grades 3 and greater organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to the underlying malignancy and occurring within 30 days of study cell infusion and does not resolve within 72 hours. Treatment-related death within 8 weeks of the study cell infusion.
Time Frame: Within 30 days of study cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
Number analyzed (Participants) | 1 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 53 days for the Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) Arm/Group, and 1 year and 4 months for the Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2) Arm/Group.
Arm/Group | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2)
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) (N=1) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2) (N=2)
Edema: head and neck (General disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Syndromes - Other (Specify, hemophagocytic syndrome) (Immune system disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-MAGE-A3 A1 TCR PBL 1x10^9 Cells + Interleukin-2 (IL-2) (N=1) | Anti-MAGE-A3 A1 TCR PBL 1x10^8 Cells + Interleukin-2 (IL-2) (N=2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0)
Fibrinogen (Investigations) | 1 (1) | 0 (0)
Hemoglobin (Investigations) | 1 (1) | 2 (2)
Ileus, GI (functional obstruction of bowel, i.e., neuro-constipation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Leukocytes (total WBC) (Investigations) | 1 (1) | 0 (0)
Lymphopenia (Investigations) | 1 (1) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1) | 2 (2)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1) | 1 (1)
Platelets (Investigations) | 1 (1) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02153905/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT02153905/ICF_001.pdf